CLINICAL TRIAL: NCT02931604
Title: Pilot Study Designed to Clinically Evaluate Sinus Wash Device Prototypes in Patients With Sinusitis During Endoscopic Sinus Surgery (ESS) and in the Hospital Outpatient
Brief Title: Study Designed to Clinically Evaluate Sinus Wash Device Prototypes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SinuSafe Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNS001
Record Dates: First submitted 2016-09-13; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Sinusitis; Maxillary Sinusitis
Keywords: sinus wash; sinus lavage; Sinusitis
MeSH Terms: conditions — Sinusitis; Maxillary Sinusitis

ARMS (1):
- Sinus irrigation (Experimental): Sinus irrigation intervention
  Interventions: Device: SinuSafe Medical Device for Maxillary Sinus

INTERVENTIONS:
Device: SinuSafe Medical Device for Maxillary Sinus — Sinus lavage via the natural sinus ostium, without ostial dilation.

SUMMARY:
The purpose of this study is to clinically evaluate sinus wash device prototypes in patients with sinusitis during Endoscopic Sinus Surgery (ESS) and in the hospital outpatient

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-65 years of age.
2. Signs and symptoms of acute exacerbation during chronic maxillary sinusitis.
3. Pain higher than 5 in VAS of 0-10.
4. Able to understand and provide written informed consent.

Exclusion Criteria:

1. Patients who have a clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation as determined by medical history based on the opinion of the investigator.
2. Extensive sinonasal polyps that may interfere with the treatment procedure.
3. Previous sinonasal surgery.
4. Acute exacerbation of sinusitis in the frontal or sphenoid sinuses.
5. Sinonasal osteoneogenesis.
6. Cystic fibrosis.
7. Sinonasal tumors or obstructive lesions.
8. Presence of features consistent with sinus fungal disease on CT or physical examination.
9. History of facial trauma that distorted the sinus anatomy.
10. Ciliary dysfunction.
11. History of insulin dependent diabetes.
12. Not able to stop anti-coagulant (e.g., warfarin) until the International Normalized Ratio (INR) is below 1.5.
13. Not able to stop anti-platelet (e.g., clopidogrel, aspirin, etc.) for at least 14 days prior to study procedure.
14. Not able to stop any non-steroidal anti-inflammatory medications and homeopathic medications for at least 14 days prior to the study procedure.
15. Pregnancy.
16. Psychiatric disease.
17. Currently participating in other drug or device studies.
18. Investigator's opinion that the subject should not be in the study such as any conditions that could compromise the wellbeing of the patient or integrity of the study or prevent the patient from meeting or performing study requirements.
19. Patient is not capable of following the study schedule for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-11 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Within day 1
  Presence of adverse events

SECONDARY OUTCOMES:
Mucosal damage visual inspection | Within 1 hour
  Visual inspection of sinus mucosa with the endoscope looking for mucosal damage.
Syringe visual inspection | Within 1 hour
  Visual inspection of the aspirated liquids looking for bleeding. Excess nasal bleeding shall be defined as a doctor decision to use sinus or nasal packing.
Pain during procedure | Within 1 hour
  Pain during procedure with the VAS pain scale
Usability & Tolerability Questionnaire | Within 1 hour
  Usability & Tolerability Questionnaire
Mucus leftovers visual inspection | Within 1 hour
  Visual inspection of sinus mucosa with the endoscope looking for mucus leftovers
Mucus aspiration into the syringe | Within 1 hour
  Mucus aspiration into the syringe (yes/ no and time)
Pain relief | Within 1 hour
  Pain relief in the post-treatment VAS pain scale
Time measurements of cannula insertion. | Within 1 hour
  Time measurements of cannula insertion
Time measurements of irrigation and aspiration | Within 1 hour
  Time measurements of irrigation and aspiration
SNOT 20 questionnaire | Within 1 hour
  SNOT 20 questionnaire (Hebrew version) to evaluate the patient's severity level before the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Itzhak Braverman, Professor, Principal Investigator — Hillel Yaffe Medical Center